CLINICAL TRIAL: NCT06287164
Title: Optimization of Therapy in the Italian Management of Heart Failure: OPTIMA-HF Observational Study
Brief Title: Management of Heart Failure in Italian Outpatients Clinics: Observational Study
Acronym: OPTIMA-HF
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: 101
Record Dates: First submitted 2024-02-20; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection on heart failure therapy and follow up

SUMMARY:
OPTIMA-HF is an observational, cross-sectional, multicenter, real-life study conducted in two different clinical settings: HF outpatients' clinics of Italian University Hospitals and territorial Cardiology outpatients' services.

Aim of the Optimization of Therapy in the Italian Management of Heart Failure [OpTIMa-HF] Registry is to collect data on HF patients followed in different Italian outpatients' settings to describe the current Italian population of HF patients, in terms of demographic characteristics and disease features, with a specific focus on guideline-directed medical therapy (GDMT) prescription, assessing its improvement after educational activities. In the present analysis we report the baseline data on the general enrolled population with a specific focus on HFrEF treatment adherence and prescription rates, according to the most recent European Guidelines.

ELIGIBILITY:
Inclusion Criteria: age >18 years, post-menopausal, permanent sterile, or childbearing potential on highly effective contraceptive methods women, stable clinical conditions (NYHA class I-III), outpatients setting, capability to understand the study procedures and sign the informed consent form.

Exclusion Criteria: any clinical condition that would have jeopardized patient safety while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients in stable clinical conditions
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
HF treatment adherence according to the most recent European Guidelines | 12 months
  Outpatients clinic treatment adherence will be measured as the percentage of patients receiving guideline-directed medical therapy prescriptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No